CLINICAL TRIAL: NCT00004136
Title: A Phase II Study of Radiofrequency Ablation of Unresectable Liver Tumors
Brief Title: Heat Therapy in Treating Patients With Unresectable Primary or Metastatic Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID97-328; P30CA016672 (NIH); MDA-ID-97328 (Other: UT MD Anderson Cancer Center); NCI-G99-1613; CDR0000067366 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-12-10; First posted 2004-08-20 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Liver Cancer; Metastatic Cancer
Keywords: stage III childhood liver cancer; stage IV childhood liver cancer; recurrent childhood liver cancer; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; liver metastases
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis; Carcinoma, Hepatocellular | interventions — Radiofrequency Ablation; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heat Therapy (Experimental)
  Interventions: Procedure: Radiofrequency Ablation

INTERVENTIONS:
Procedure: Radiofrequency Ablation — Tumors heated to target temperature by electrodes for maximum of 20 minutes
  Other Names: Heat Therapy

SUMMARY:
RATIONALE: Heating tumors to several degrees above body temperature may kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of heat therapy in treating patients who have unresectable primary or metastatic liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of radiofrequency ablation in patients with primary or metastatic liver cancer. II. Determine disease free survival, local recurrence rate in treated lesions as compared to known recurrence rates after hepatic cryoablation, and overall survival in this patient population receiving this regimen.

OUTLINE: Patients undergo laparoscopic or open laparotomy surgical procedure to identify unresectable tumors by ultrasound. Tumors are heated to a target temperature by electrodes for a maximum of 20 minutes. To achieve a 1 cm margin of ablated tissue around each lesion, multiple ablation courses may be performed, depending on the size of the lesions and the time required to complete the treatment. Patients may be retreated if tumor recurs or new disease appears. Patients are followed at 1 month, every 3 months for the first 2 years, every 6 months for next 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 59 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of unresectable malignant primary or metastatic liver tumors Tumors are deemed unresectable based on the following factors: 1-10 liver tumors Bilobar liver tumors Location of 1 or more lesions near a major intrahepatic vascular structure (hepatic vein, portal vein, vena cava) Severe cirrhosis to preclude a major liver resection No unresectable extrahepatic disease Prior failure of other therapeutic modalities allowed No more than moderate ascites No hepatic encephalopathy

PATIENT CHARACTERISTICS: Age: Any age Performance status: Zubrod 0-1 Life expectancy: At least 3 months Hematopoietic: Not specified Hepatic: No severe liver dysfunction (Child's Class C) Bilirubin no greater than 3.0 mg/dL Albumin no greater than 3.0 mg/dL PT no greater than 50% above normal Renal: No renal dysfunction Creatinine less than 2.0 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No altered mental status No active infection

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 1998-03-09 (Actual); Primary Completion 2006-01-25 (Actual); Study Completion 2006-01-25 (Actual)

PRIMARY OUTCOMES:
Efficacy of Radiofrequency Ablation in Patients with Primary or Metastatic Liver Cancer | 1 Month

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Curley, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org